CLINICAL TRIAL: NCT02549586
Title: Autologous Hematopoietic Stem Cell Transplantation for Allogeneic Organ Transplant Tolerance
Acronym: ASCOTT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary A Levy, O. Ont. MD. FRCP AGAF (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Gary A Levy, O. Ont. MD. FRCP AGAF, Gary A Levy, O. Ont. MD. FRCP AGAF, University of Toronto
Organization: University of Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tol 001
Record Dates: First submitted 2015-09-01; First posted 2015-09-15 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Complication of Transplanted Organ, Nos
Keywords: solid organ transplant; immune tolerance; autologous stem cell transplant; blood and marrow transplant; autoimmune disease
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Pt are receiving everolimus in combination with autologous stem cell transplant to induce tolerance
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous HSCT (Experimental): Eligible participants will undergo an Autologous Hematopoietic Stem Cell Transplant (HSCT) as a two-step intervention.
  Interventions: Drug: Autologous Hematopoietic Stem Cell Transplant

INTERVENTIONS:
Drug: Autologous Hematopoietic Stem Cell Transplant — Step 1: Participants will receive intravenous chemotherapy and cytokine-based treatment for mobilization of hematopoietic stem cells (HSC) into the circulation, followed by collection using peripheral vein leukopheresis. The HSC graft product will undergo ex vivo purification with CD34 selection using Miltenyil CliniMACS and cryopreserved.
  Step 2: Intravenous busulphan, cyclophosphamide and anti-thymocyte globulin will be administered to participants to achieve immune ablation prior to the infusion of the participants' own thawed HSC graft product (HSC transplant). Routine supportive measures will be employed during the recovery from the chemotherapy and HSCT. Participants' immune suppression will be stopped at the time of immunoablative therapy and will be switched to everolimus which will be discontinued at 6 months post HSCT.
  Other Names: HSCT

SUMMARY:
This open-label, proof-of-principle two center cohort study will evaluate the ability of autologous hematopoietic stem cell transplantation to induce tolerance in recipients of deceased or live donor liver transplants (ASCOTT). A maximum of 10 participants will be entered at a minimum of 3 months post liver transplant. The participants will undergo autologous hematopoietic stem cell transplants (HSCT) to "re-educate" their immune systems to accept the graft without the need for long term immunosuppression (tolerance).

DETAILED DESCRIPTION:
Although short-term results for liver transplantation are excellent, the need for immunosuppression limits quality of life and long-term survival.

Investigators plan to examine the utility and safety of autologous hematopoietic stem cell transplantation (HSCT) to allow withdrawal of immunosuppression in 10 liver transplant recipients who are at a high risk of developing recurrent liver damage from repeated bouts of rejection, or recurrent disease or who have a high likelihood of developing serious medical complications from complications of immune suppression.

Hematopoietic stem cells will be mobilized, purified and cryopreserved. Following a chemotherapy and Anti-thymocyte Globulin (ATG) based-regimen for immune ablation, the purified stem cells will be thawed and infused back into participants (autologous hematopoietic stem cell transplant - HSCT). Participants will be converted to everolimus, a mammalian target of rapamycin inhibitor (mTORi), which will be continued for 6 months and then withdrawn based on histologic evidence of graft acceptance.

Participants will be followed closely for a total of 24 months for any biochemical and histologic evidence of tolerance or rejection. Re-vaccination to common viral and bacterial antigens will be undertaken as required using a standard protocol for recipients of a hematopoietic stem cell transplant (HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years of age or older.
2. Participants must be a minimum of 6 months post-transplant;
3. Participants are recipients of a hepatic allograft for alcohol induced liver disease; or a genetic form of liver disease such as hemochromatosis or Wilson's disease; or an autoimmune liver disease including sclerosing cholangitis, autoimmune hepatitis, and/or primary biliary cirrhosis.
4. Participants have a complication of transplantation that might be ameliorated by HSCT and/or withdrawal of immunosuppression such as: evidence of recurrent autoimmune disease in the graft; repeated episodes (minimum of 2) of acute cellular rejection; and/ or development of adverse events related to immune suppression which have not been well managed by conventional methods including drug dose reduction or substitution of other medications. Examples include progression of renal dysfunction, repeated infections, neurologic complications, cardiovascular complications, or post-transplant lymphoproliferative disease (PTLD) that has been in remission for at least 12 months. These complications must be deemed serious enough to warrant inclusion in the study by the investigator.

Exclusion Criteria:

1. Participants < 18 yr.
2. Participants with cardiac, renal, pulmonary, hepatic, or other organ impairment that would limit their ability to receive dose intensive chemotherapy;
3. Participants with any active or chronic infection. Participants with previous reactivation of Epstein-Barr virus, cytomegalovirus , BK, human herpesvirus 6 or varicella-zoster virus would be considered eligible if the virus has returned to a latent state;
4. Participants who are seropositive for HIV1, HIV2, Hepatitis B Surface Antigen, and Hepatitis C;
5. Participants with a previous history of a malignancy other than squamous or basal cell carcinoma of the skin, or post-transplant lymphoproliferative disease (PTLD);
6. Participants whose life expectancy is severely limited by another co-morbid illness;
7. Participants with evidence of myelodysplasia, other non-autoimmune cytopenia, or an inherited immunodeficiency state;
8. Pregnancy or Participants who are unwilling to practice two active forms of contraception during the time of chemotherapy administration. Participants must be willing to commit to not becoming pregnant from enrollment in the study until 2 years following their HSCT.
9. Participants unable to comply with the medical treatment specified in the protocol;
10. Participants unable to give written informed consent in accordance with research ethics board guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop tolerance post autologous HSCT | 24 months post HSCT
  Number of patients who develop tolerance at 24 months post HSCT as defined clinically and histologically in the absence of any immunosuppression in liver transplant recipients.

SECONDARY OUTCOMES:
HSCT mortality | 2 years post HSCT
HSCT related morbidity | at 2 years post HSCT
Rate of immune reconstitution | at 2 years post HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Levy, MD FRCP AGAF, Principal Investigator — University of Toronto Transplant Institute - Multi Organ Transplant Program; Harold L Atkins, MD FRCP(C), Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hopital, Ottawa, Ontario
  - Multi-Organ Transplant Program, Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Sykes M, Levy G. Advances in transplantation. Semin Immunol. 2011 Aug;23(4):222-3. doi: 10.1016/j.smim.2011.08.013. Epub 2011 Sep 22. No abstract available. PMID 21943504
- [Background] Sayegh MH, Carpenter CB. Transplantation 50 years later--progress, challenges, and promises. N Engl J Med. 2004 Dec 23;351(26):2761-6. doi: 10.1056/NEJMon043418. No abstract available. PMID 15616214
- [Background] Azzi JR, Sayegh MH, Mallat SG. Calcineurin inhibitors: 40 years later, can't live without .. J Immunol. 2013 Dec 15;191(12):5785-91. doi: 10.4049/jimmunol.1390055. PMID 24319282
- [Background] Selzner N, Grant DR, Shalev I, Levy GA. The immunosuppressive pipeline: meeting unmet needs in liver transplantation. Liver Transpl. 2010 Dec;16(12):1359-72. doi: 10.1002/lt.22193. PMID 21117245
- [Background] Kaplan B, Qazi Y, Wellen JR. Strategies for the management of adverse events associated with mTOR inhibitors. Transplant Rev (Orlando). 2014 Jul;28(3):126-33. doi: 10.1016/j.trre.2014.03.002. Epub 2014 Mar 12. PMID 24685370
- [Background] Gotthardt DN, Bruns H, Weiss KH, Schemmer P. Current strategies for immunosuppression following liver transplantation. Langenbecks Arch Surg. 2014 Dec;399(8):981-8. doi: 10.1007/s00423-014-1191-9. Epub 2014 Apr 20. PMID 24748543
- [Background] Sachs DH, Kawai T, Sykes M. Induction of tolerance through mixed chimerism. Cold Spring Harb Perspect Med. 2014 Jan 1;4(1):a015529. doi: 10.1101/cshperspect.a015529. PMID 24384815
- [Background] Kawai T, Sachs DH, Sykes M, Cosimi AB; Immune Tolerance Network. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2013 May 9;368(19):1850-2. doi: 10.1056/NEJMc1213779. No abstract available. PMID 23656665
- [Background] Xie L, Ichimaru N, Morita M, Chen J, Zhu P, Wang J, Urbanellis P, Shalev I, Nagao S, Sugioka A, Zhong L, Nonomura N, Takahara S, Levy GA, Li XK. Identification of a novel biomarker gene set with sensitivity and specificity for distinguishing between allograft rejection and tolerance. Liver Transpl. 2012 Apr;18(4):444-54. doi: 10.1002/lt.22480. PMID 22162188
- [Derived] Chruscinski A, Juvet S, Moshkelgosha S, Renner E, Lilly L, Selzner N, Bredeson C, Grant D, Adeyi O, Fischer S, Demetris AJ, Zhang J, Epstein M, Macarthur M, Clement AM, Khalili K, Allan D, Altouri S, Bence-Bruckler I, Cattral M, Fulcher J, Galvin Z, Ghanekar A, Greig P, Huebsch L, Humar A, Kew A, Kekre N, Kim TK, McDiarmid S, Martin L, McGilvray I, Sabloff M, Sapisochin G, Selzner M, Smith R, Tinckam K, Yi TJ, Levy G, Atkins H. Autologous Hematopoietic Stem Cell Transplantation for Liver Transplant Recipients With Recurrent Primary Sclerosing Cholangitis: A Pilot Study. Transplantation. 2022 Mar 1;106(3):562-574. doi: 10.1097/TP.0000000000003829. PMID 34049362